CLINICAL TRIAL: NCT01691872
Title: An Open-label, Single Centre, Parallel Group Study to Evaluate the Safety and Pharmacokinetics of Single Oral Doses of Retigabine Extended Release (XR) Formulation in Healthy Adult Japanese and Caucasian Subjects
Brief Title: Pharmacokinetic Study of Retigabine Extended Release (XR) Formulation in Healthy Adult Japanese and Caucasian Subjects
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Development plan of retigabine XR in Japan was readjusted.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 116247
Record Dates: First submitted 2012-09-13; First posted 2012-09-25 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Epilepsy, Partial
MeSH Terms: conditions — Epilepsies, Partial | interventions — ezogabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Japanese (Experimental): Retigabine 300mg single-dose
  Interventions: Drug: Retigabine
- Caucasian (Experimental): Retigabine 300mg single-dose
  Interventions: Drug: Retigabine

INTERVENTIONS:
Drug: Retigabine — Retigabine

SUMMARY:
This is an open-label, single centre, parallel group study to evaluate the safety and pharmacokinetics of single oral doses of retigabine XR formulation in healthy adult Japanese subjects. To compare the pharmacokinetic and safety profile, Caucasian subjects are also incorporated. This study is intended to facilitate inclusion of Japanese patients in the global phase III program for retigabine XR formulation.

ELIGIBILITY:
Inclusion Criteria:

* Male subject between 20 and 45 years of age inclusive, at the time of signing the informed consent.
* Japanese ancestry defined as being born in Japan, having four ethnic Japanese grandparents, holding a Japanese passport or identity papers and being able to speak Japanese. OR Caucasian defined as an individual having four grandparents who are all descendents of the original people of Europe.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and 12-lead ECG. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight ≥ 50 kg and BMI within the range 18.5 - 24.9 kg/m2 (inclusive).
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed separately. This criterion must be followed from the time of the first dose of study medication until 1 week post-last dose
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* AST, ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Single QTcB or QTcF< 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.

Exclusion Criteria:

* Subject has made a suicide attempt in the past or, in the investigator's judgment, poses a significant suicide risk. Evidence of serious suicide risk may include any history of suicidal behavior in the past 6 months and/or any suicidal ideation of type 4 or 5 on the Columbia Suicide Severity Rating Scale (C-SSRS).
* A positive pre-study Hepatitis B surface antigen, Hepatitis C antibody or HIV antigen/antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 360 ml of beer, 150 ml of table wine or 45 ml of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Unable to refrain from consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10-10 (Actual); Primary Completion 2012-10-18 (Actual); Study Completion 2012-10-18 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ of retigabine | up to 96h post dose
  Area under the concentration-time curve from pre-dose to last time of quantifiable concentration of retigabine
Cmax of retigabine | up to 96h post dose
  Maximum observed concentration of retigabine
Tmax of retigabine | up to 96h post dose
  Time of occurance of Cmax of retigabine
t1/2 of retigabine | up to 96h post dose
  Terminal phase half-life of retigabine
Adverse Events | up to 96h post dose
  Number of participants with adverse events as a measure of safety and tolerability (evaluated by the result of Clinical safety laboratory tests, vital signs, 12-lead ECG, telemetry and clinical monitoring/observation

SECONDARY OUTCOMES:
AUC0-∞ of NAMR | up to 96h post dose
  Area under the concentration-time curve from pre-dose to last time of quantifiable concentration of NAMR
Cmax of NAMR | up to 96h post dose
  Maximum observed concentration of NAMR
Tmax of NAMR | up to 96h post dose
  Time of occurance of Cmax of NAMR
t1/2 of NAMR | up to 96h post dose
  Terminal phase half-life of NAMR
fe | up to 96h post dose
  Percent of retigabine and NAMR excreted in urine
CLr | up to 96h post dose
  Renal clearance of retigabine and NAMR

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Kagoshima, Japan